CLINICAL TRIAL: NCT01511185
Title: NNC 90-1170 Mechanism of Action: A Double-blind, Randomized, Single-center, Placebo Controlled, Crossover Study to Examine Beta-cell Responsiveness to Graded Glucose Infusion in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide on the Beta-cell Responsiveness in Subjects With Type 2 Diabetes Compared to a Healthy Control Group
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-2063
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: liraglutide; Drug: placebo
- Healthy (No Intervention)

INTERVENTIONS:
Drug: liraglutide — A single dose of 7.5 mcg/kg administered subcutaneously in random order
  Other Names: NNC 90-1170
  Arms: NNC 90-1170; Placebo
Drug: placebo — A single dose administered subcutaneously in random order
  Arms: NNC 90-1170; Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to assess the effect of NNC 90-1170 on beta-cell responsiveness to increasing blood glucose concentrations in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes, either newly diagnosed with at least 2 months of diet or on OAD monotherapy for at least 3 months
* Body Mass Index (BMI): 24-35 kg/m^2 inclusive

Exclusion Criteria:

* SUBJECTS WITH TYPE 2 DIABETES
* Receipt of any investigational drug within three months prior to this trial
* Recurrent severe hypoglycemia as judged by the investigator
* Cardiac disease
* Use of any drug (except an OAD (oral anti-diabetic drug)) that in the investigator's opinion could interfere with the blood glucose level
* Haemoglobin maximum 10 g/L
* HbA1c above 12%
* Loss of more than 400 mL blood during the 3 months prior to trial start
* HEALTHY SUBJECTS
* Receipt of any investigational drug within 3 months prior to this trial
* Clinically relevant cardiac disease or any clinically significant abnormal ECG (electrocardiogram)
* Use of any drug that in the investigator's opinion could interfere with the blood glucose level
* Haemoglobin max. 10 g/L
* HbA1c at least 6%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-02; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) of Insulin Secretion Rate (ISR) over the 90-216 mg/dL glucose interval

SECONDARY OUTCOMES:
Slope of the mean ISR vs mean glucose
AUC (area under the curve) of glucagon concentration over the 90-216 mg/dL glucose interval
Insulin Clearance
NNC 90-1 170 plasma concentration
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Chang AM, Jakobsen G, Sturis J, Smith MJ, Bloem CJ, An B, Galecki A, Halter JB. The GLP-1 derivative NN2211 restores beta-cell sensitivity to glucose in type 2 diabetic patients after a single dose. Diabetes. 2003 Jul;52(7):1786-91. doi: 10.2337/diabetes.52.7.1786. PMID 12829647
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com